CLINICAL TRIAL: NCT07161284
Title: Impact of Mental Health First Aid-trained Peers on the Mental Well-being of First-year Medical Residents.
Acronym: PS-MHFA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL25_0576
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Mental Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed (Experimental): Medical residents entering their first year of specialized studies (DES) on November 1, 2025, in the city of Lyon, France.
  Interventions: Other: Exposition to trained peer-support registrars for a year
- Not exposed (No Intervention): Medical residents entering their second year of specialized studies (DES) on November 1, 2025, in the city of Lyon, France.

INTERVENTIONS:
Other: Exposition to trained peer-support registrars for a year — Exposition to trained peer-support registrars for a year
  Arms: Exposed

SUMMARY:
Medical students, especially those in postgraduate training, face a complex array of challenges such as fatigue; work-life balance conflicts; difficulties managing dual hierarchies (hospital and university). Surprisingly, residents receive little to no dedicated training in recognizing and managing psychiatric disorders, except for psychiatry residents. This gap is exacerbated by persistent stigma towards psychiatric conditions. The Mental Health First Aid (MHFA) training approach could offer an innovative solution, addressing the root of the problem. This prospective, single-center cohort study aims to compare (1) the mental well-being of first-year specialty residents in the Lyon subdivision exposed to MHFA-trained peers; with (2) the mental well-being of unexposed second-year specialty residents. The hypothesis is that exposure to peers trained in MHFA improves well-being and reduces symptoms of burnout, depression, and anxiety at 3, 6, 9, and 12 months among peer residents.

ELIGIBILITY:
Inclusion Criteria:

* subject to the non-opposition of the residents, all medical residents entering their first and second year of specialized studies (DES) on November 1, 2025, in the city of Lyon will be included in the study.

Exclusion Criteria:

* refusal to participate AND in the unlikely cases where:
* subject under guardianship or curatorship;
* subject unable to give free and informed consent;
* subject under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Well-being | Measured at Month 12
  As measured by the total score on the WEMWBS (Warwick-Edinburgh Mental Well-being Scale), a self-questionnaire. 5 point Likert scale (1-4); 14 questions

SECONDARY OUTCOMES:
Well-being | Measured at baseline, Month 3, Month 6 and Month 9
  As measured by the total score on the WEMWBS (Warwick-Edinburgh Mental Well-being Scale), a self-questionnaire. 5 point Likert scale (1-4); 14 questions
Anxiety | Measured at baseline, Month 3, Month 6, Month 9, Month 12
  As measured by anxiety subscore of the HAD (Hospital Anxiety and Depression scale), a self-questionnaire. 4 point Likert scale (0-3); 7 questions
Depression | Measured at baseline, Month 3, Month 6, Month 9, Month 12
  As measured by depression subscore of the HAD (Hospital Anxiety and Depression scale), a self-questionnaire. 4 point Likert scale (0-3); 7 questions
Burn-out | Measured at baseline, Month 3, Month 6, Month 9, Month 12
  As measured by the MBI (Maslach Burnout Inventory), a self-questionnaire. 7 point Likert scale (0-6); 22 questions.
Impact on well-being according to gender | Measured at baseline, Month 3, Month 6, Month 9, Month 12
  Differentiated impact on well-being according to gender measured by the total score on the WEMWBS (Warwick-Edinburgh Mental Well-being Scale, a self-questionnaire. 5 point Likert scale (1-4); 14 questions), analyzed via Group x Gender interaction effect.
Impact on well-being according to speciality | Measured at baseline, Month 3, Month 6, Month 9, Month 12
  Differentiated impact on well-being according to speciality measured by the total score on the WEMWBS (Warwick-Edinburgh Mental Well-being Scale, a self-questionnaire. 5 point Likert scale (1-4); 14 questions), analyzed via Group x Speciality interaction effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Urgences Psychiatriques Hôpital Edouard Herriot, GH Centre, Lyon, France, France